CLINICAL TRIAL: NCT01329094
Title: Physical Activity in Patients With Severe Mental Illness
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Lene Nyboe Jacobsen, Aarhus University
Other Study IDs: Lene Nyboe Jacobsen 2
Record Dates: First submitted 2010-08-09; First posted 2011-04-05 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-04

CONDITIONS: Mental Disorders
Keywords: Severe mental illness; physical activity; evaluation
MeSH Terms: conditions — Mental Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with severe mental illness: In-patients and out-patients with severe mental illness attending treatment at Aarhus University Hospital, Risskov.
- Healthy controls: Healthy controls recruited from staff members at Aarhus University Hospital, Risskov

SUMMARY:
The aim of the study was to evaluate the applicability of the Physical Activity Scale (PAS) in relation to patients with severe mental illness. The study hypothesised that physical activity levels among patients with severe mental illness was significantly lower than healthy controls. The physical activity level of patients with severe mental illness attending Aarhus University Hospital, Risskov in comparisons with healthy controls matched on gender and age was assessed with PAS.

DETAILED DESCRIPTION:
The study population of interest was psychiatric in- or outpatients from Aarhus University Hospital , Risskov, some of whom were referred for physiotherapeutic treatment. The patients were compared with healthy controls matched on gender and age, recruited from hospital staff including administrative employees.Patients and controls were included in the study after giving informed consent, according to the Declaration of Helsinki 2008. All participants assessed their physical activity level by completing the PAS questionnaire twice within a time period of 5-7 days for evaluation of the test-retest reliability of PAS. For patients, PAS was administered as an interview, and for controls as a self-questionnaire. Several physiotherapists (PTs) were involved in interviewing the patients.

In total, 47 hospitalized patients or outpatients and 28 controls were included in the study. In comparison with controls, the physical activity level of daily life of the patients was statistically significantly lower, even though the average physical activity level of the healthy controls was just above 'moderate physical activity'.

There was a satisfactory test-retest reliability of PAS when applied to both mentally ill patients and healthy controls. PAS was found to be an applicable method for evaluating physical activity levels in patients with severe mental illness, and also useful in measuring changes in physical activity levels.

ELIGIBILITY:
Inclusion Criteria:

* All in and outpatients attending psychiatric treatment at Aarhus University Hospital, Risskov

Exclusion Criteria:

* Physical disablement, subject to coercive treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Psychiatric in- and outpatients admitted to Aarhus University Hospital, Risskov, Denmark
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Physical activity level | The average physical activity level of the past week is assessed (one week)
  The physical activity level is assessed using the Physical Activity Scale, which is based ion the concept that the intensity of physical activity can be expressed in metabolic equivalents.

CONTACTS AND LOCATIONS:
Overall Officials: Lene N Jacobsen, PT, Msc, Principal Investigator — Aarhus University, Risskov